CLINICAL TRIAL: NCT05098678
Title: The Effects of Zinc Gluconate Supplementation on Several Genes Expression, the Serum Level of Inflammatory Factors, Quality of Life, and Disease Activity in Patients With Behcet Syndrome: Double-blind Randomized Controlled Clinical Trial
Brief Title: Zinc Supplementation and Behçet's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Beitullah Alipour, Beitullah Alipour, Ph.D., Prof., Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64693
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc gluconate (Experimental): zinc gluconate tablet daily (120 mg each tablet containing 30 mg elemental zinc)
  Interventions: Dietary Supplement: Zinc gluconate
- Control (Placebo Comparator): Placebo (microcrystalline cellulose): 1 tablet (120 mg each)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — 120 mg each tablet containing 30 mg elemental zinc
  Arms: Zinc gluconate
Dietary Supplement: Placebo — Placebo (microcrystalline cellulose): 1 tablet (120 mg each)
  Arms: Control

SUMMARY:
To study the effects of zinc gluconate supplementation on patients with Behçet's syndrome, 50 patients will be randomly allocated to two groups: placebo group or zinc group (one tablet of 30 mg/day elemental zinc) for 12 weeks. All participants will be asked not to alter their diet, medication, and physical activity during the study. At the first and the end of the intervention, genes and proteins expression, the serum level of inflammatory factors, quality of life, disease activity, anthropometric measures, physical activity and serum level of zinc will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20 to 50 years (premenopausal woman)
* Diagnosis of Behcet's disease by a rheumatologist according to IBCD (The International Criteria for Behcet's Disease)
* Patients who want to participate in the study

Exclusion Criteria:

* Pregnancy and lactation
* History of diabetes and other chronic diseases
* Smoking and alcohol consumption over the past year
* History of other autoimmune diseases
* Consumption of nutritional and antioxidant supplements over two months prior to the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Toll-like Receptor-2 gene expression | 12 weeks
  2-ΔΔCT
Toll-like Receptor-4 gene expression | 12 weeks
  2-ΔΔCT
Toll-like Receptor-2 protein expression | 12 weeks
  The mean fluorescence intensity
Toll-like Receptor-4 protein expression | 12 weeks
  The mean fluorescence intensity
Serum level of tumor necrosis factor-alpha | 12 weeks
  pg/ml
NLRP3 gene expression | 12 weeks
  2-ΔΔCT
Caspase-1 gene expression | 12 weeks
  2-ΔΔCT
Serum level of interleukin-1 beta | 12 weeks
  pg/ml
Serum level of zinc | 12 weeks
  ug/dl

SECONDARY OUTCOMES:
Behçet's disease quality-of-life | 12 weeks
  Behçet's disease quality-of-life. The score ranged between 0-30. Zero means high quality of life and 30 means low quality of life.
Disease activity | 12 weeks
  Behcets Disease Activity

CONTACTS AND LOCATIONS:
Locations (1):
- Tabriz University of Medical Sciences, Tabriz, East Azerbaijan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faghfouri AH, Khabbazi A, Baradaran B, Khajebishak Y, Baghbani E, Noorolyai S, Rahmani S, Seyyed Shoura SM, Alipour M, Alipour B. Immunomodulatory and clinical responses to zinc gluconate supplementation in patients with Behcet's disease: A double-blind, randomized placebo-controlled clinical trial. Clin Nutr. 2022 May;41(5):1083-1092. doi: 10.1016/j.clnu.2022.03.019. Epub 2022 Mar 30. PMID 35413570